CLINICAL TRIAL: NCT05591209
Title: Pattern of Admission and Outcome of Patients Admitted to the Intensive Care Unit of a Tertiary Hospital in Low Resource Setting. A Cohort Study
Brief Title: Pattern of Admission and Outcome of Patients Admitted to the Intensive Care
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Haramaya Unversity (Other)
Responsible Party: Principal Investigator, Badhaasaa, Dr, Haramaya Unversity
Other Study IDs: IHRERC/052/2022
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Failure; Treatment Outcome
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alive and Dead: Following ICU admission patients are followed until discharge with the outcome of alive or dead

SUMMARY:
The study was a retrospective observational cohort where patient medical record review was done and data were gathered on 419 cases. The ICU admission pattern and patient outcome were the primary outcomes presented in the manuscript.

DETAILED DESCRIPTION:
The study was conducted at a teaching University hospital in a low-resource setting retrospectively on admission to ICU over the last five years. samples were selected using a simple random sampling technique to come up with the desired number.

ELIGIBILITY:
Inclusion Criteria:

* complete medical record
* admission to ICU

Exclusion Criteria:

* patients who were transferred or self discharged

Ages: 4 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients admitted to ICU of HrU- HFCSH
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
pattern of admission and outcome of patients admitted to the Intensive care Unit of a tertiary hospital in Low resource setting. A cohort study | 1 month
  a retrospective cohort study

CONTACTS AND LOCATIONS:
Locations (2):
- Ethiopia (2):
  - HFSUH, Harar, Harari NS
  - Haramaya university, Harar

IPD SHARING:
Plan to Share IPD: No
IPD will not be exposed